CLINICAL TRIAL: NCT07274969
Title: The Effect of Caffeine Therapy in Cardiovascular Stability in Preterm Neonates: a Prospective Study at the Neonatal Intensive Care Unit of Assiut University Children Hospital
Brief Title: The Effect of Caffeine Therapy in Cardiovascular Stability in Preterm Neonates at Assiut University Children Hospital NICU
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Margret Azer, Resident at Pediatric Department, Assiut University, Assiut University
Other Study IDs: caffeine therapy
Record Dates: First submitted 2025-09-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Preterm Neonates; Apnea of Prematurity
Keywords: Preterm neonates; apnea of prematurity
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm neonates: Preterm neonates receiving standard caffeine citrate therapy for apnea of prematurity, including a loading dose of 20-25 mg/kg followed by maintenance dosing (5-10 mg/kg daily). Cardiovascular parameters and side effects are monitored longitudinally.

SUMMARY:
Preterm neonates younger than 37 weeks gestational age receiving caffeine therapy for apnea of prematurity in a NICU setting.

DETAILED DESCRIPTION:
The study population consists of 40 preterm neonates admitted to the Neonatal Intensive Care Unit at Assiut University Children Hospital. Inclusion criteria restrict participants to those with a gestational age below 37 weeks who are prescribed caffeine citrate therapy to manage apnea of prematurity. Neonates with major congenital anomalies or those requiring vasopressors at baseline are excluded. The cohort is monitored closely for cardiovascular parameters and adverse reactions related to caffeine administration. Demographic and clinical baseline data include prenatal risk factors, gestational and postnatal age, and birth weight. This focused population allows investigation of caffeine's impact on vulnerable cardiovascular physiology during early neonatal life.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age <37 weeks
* Receiving caffeine therapy for apnea of prematurity
* Hemodynamically stable before caffeine initiation

Exclusion Criteria:

* Presence of major congenital anomalies
* Use of vasopressors at baseline
* Severe intraventricular hemorrhage (Grade III-IV)

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates receiving standard caffeine citrate therapy for apnea of prematurity, including a loading dose of 20-25 mg/kg followed by maintenance dosing (5-10 mg/kg daily). Cardiovascular parameters and side effects are monitored longitudinally.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean arterial blood pressure after caffeine therapy in preterm neonates. | Baseline before caffeine administration and at 1, 6, 12, and 24 hours after caffeine dose.
  Mean change in mean arterial blood pressure (mmHg) in preterm neonates receiving caffeine therapy for apnea of prematurity, comparing post-caffeine values with baseline pre-caffeine values.
Change in perfusion index after caffeine therapy in preterm neonates. | Baseline before caffeine administration and at 1, 6, 12, and 24 hours after caffeine dose.
  Mean change in perfusion index (unitless value from pulse oximeter) in preterm neonates receiving caffeine therapy for apnea of prematurity, comparing post-caffeine values with baseline pre-caffeine values.
Change in heart rate after caffeine therapy in preterm neonates. | Baseline before caffeine administration and at 1, 6, 12, and 24 hours after caffeine dose.
  Mean change in heart rate (beats per minute) in preterm neonates receiving caffeine therapy for apnea of prematurity, comparing post-caffeine values with baseline pre-caffeine values, and documenting episodes of tachycardia defined as heart rate greater than 180 beats per minute.